CLINICAL TRIAL: NCT03785054
Title: A Phase I, Randomised, Double-blind, Placebo Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral HTL0014242 in Healthy Adults
Brief Title: Phase 1, Healthy Subject, Safety, Tolerability and Pharmacokinetic Study of mGlu5 NAM HTL0014242
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: HTL0014242-101
Record Dates: First submitted 2018-12-13; First posted 2018-12-24 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Single ascending dose
Who Masked: Participant, Investigator
Masking Description: • Placebo capsules will be identical in appearance to the HTL0014242 capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): 6 subjects receiving a single dose of 1 mg capsule HTL0014242 and 2 subjects receiving matching placebo oral capsule
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule
- Cohort 2 (Experimental): 6 subjects receiving single dose of HTL0014242 and 2 subjects receiving matching placebo oral capsule. The dose of HTL0014242 selected in an escalating manner following review of safety and tolerability data from the previous lower dose level.
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule
- Cohort 3 (Experimental): 6 subjects receiving single dose of HTL0014242 and 2 subjects receiving matching placebo oral capsule. The dose of HTL0014242 selected in an escalating manner following review of safety and tolerability data from the previous lower dose level.
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule
- Cohort 4 (Experimental): 6 subjects receiving single dose of HTL0014242 and 2 subjects receiving matching placebo oral capsule. The dose of HTL0014242 selected in an escalating manner following review of safety and tolerability data from the previous lower dose level.
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule
- Cohort 5 (Experimental): 6 subjects receiving single dose of HTL0014242 and 2 subjects receiving matching placebo oral capsule. The dose of HTL0014242 selected in an escalating manner following review of safety and tolerability data from the previous lower dose level.
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule
- Cohort 6 (Experimental): 6 subjects receiving single dose of HTL0014242 and 2 subjects receiving matching placebo oral capsule. The dose of HTL0014242 selected in an escalating manner following review of safety and tolerability data from the previous lower dose level.
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule
- Cohort 7 (Experimental): 6 subjects receiving single dose of HTL0014242 and 2 subjects receiving matching placebo oral capsule. The dose of HTL0014242 selected in an escalating manner following review of safety and tolerability data from the previous lower dose level.
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule
- Cohort 8 (Experimental): 6 subjects receiving single dose of HTL0014242 and 2 subjects receiving matching placebo oral capsule. The dose of HTL0014242 selected in an escalating manner following review of safety and tolerability data from the previous lower dose level.
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule
- Cohort 9 (Experimental): 6 subjects receiving single dose of HTL0014242 and 2 subjects receiving matching placebo oral capsule. The dose of HTL0014242 selected in an escalating manner following review of safety and tolerability data from the previous lower dose level.
  Interventions: Drug: HTL0014242; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: HTL0014242 — HTL0014242 is a selective negative allosteric modulator (NAM) for the metabotropic glutamate (mGlu) receptor 5 subtype (mGlu5)
Drug: Placebo oral capsule — Placebo treatment

SUMMARY:
This is the first time HTL0014242 will be administered to humans. The principal aim of this study is to obtain safety and tolerability data when HTL0014242 is administered orally as single doses to healthy subjects. This information, together with the pharmacokinetics data, will help establish the doses and dosing regimen suitable for future studies in patients

DETAILED DESCRIPTION:
This study will comprise a single dose, sequential group design. Overall, up to 72 subjects will be studied in up to 9 planned groups (Groups 1 to 9), with each group consisting of 8 subjects. In addition, a further 6 subjects will participate in a crossover food effect arm.

Subjects will be screened within 28 days prior to dosing. Each subject will participate in 1 treatment period only, except the food effect arm where subjects will be dosed both fed and fasted. Subjects will reside at the clinical research unit from Day -1 (the day before dosing) to Day 5.

All subjects will return for a follow-up visit 7 to 14 days after dosing. The investigator (or designee) may also request that the subject return for an additional follow up visit.

In each of groups 1 to 9, 6 subjects will receive a single dose of HTL0014242 and 2 subjects will receive placebo oral capsule in accordance with a randomisation schedule. In the food effect arm, 6 subjects will receive a single dose of HTL0014242 in both the fed and fasted state, separated by 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females of any race, between 18 and 55 years of age, inclusive.
2. Body mass index between 18.0 and 30.0 kg/m2, inclusive, with a body weight of at least 50.0 kg.
3. In good physical and mental health, including no clinically significant findings from medical history, physical examination, psychiatric examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening or check in as assessed by the investigator (or designee).
4. Females who are not pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
5. Has clinical laboratory test results within the reference ranges of the testing laboratory, with the exception of results outside the reference ranges that are deemed not clinically significant by the Investigator (or designee) at screening and check-in.
6. Has supine blood pressure and pulse rate within the following ranges after 5 minutes rest: systolic blood pressure 90 to 140 mmHg, diastolic blood pressure 40 to 90 mmHg, and pulse rate 45 to 90 bpm.
7. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

1. Past or current history of any mental, behavioural, or neurodevelopmental disorder as defined by the tenth revision of the International Classification of Diseases (ICD-10)16 including, but not limited to, diagnoses of: organic, including symptomatic, mental disorders (F00-F09); mental and behavioural disorders due to psychoactive substance use (F10-F19); schizophrenia, schizotypal, and delusional disorders (F20-F29); mood [affective] disorders (F30-F39); neurotic, stress-related, and somatoform disorders (F40-F48); disorders of adult personality and behaviour (F60-F69).
2. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, gastrointestinal, neurological, respiratory, or endocrine disorder, as determined by the Investigator (or designee).
3. Active or history of cardiovascular or cerebrovascular disease, including hypertension, angina, ischaemic heart disease, transient ischaemic attacks, bundle branch block, evidence of myocardial ischaemia, stroke, and peripheral arterial disease sufficient to cause symptoms and/or require therapy to maintain stable status.
4. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
5. Active neoplastic disease or history of any neoplastic disease within 5 years of screening (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitely treated with standard of care).
6. Active infection (eg, sepsis, pneumonia, abscess) or a serious infection (eg, resulting in hospitalisation or requiring parenteral antibiotic treatment) within 6 weeks prior to dosing.
7. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
8. Any of the following at screening and/or predose:

   1. QT interval corrected for heart rate using Fridericia's method (QTcF) >450 ms confirmed by repeat measurement
   2. QRS duration >110 ms confirmed by repeat measurement
   3. PR interval >220 ms confirmed by repeat measurement
   4. findings which would make QTc measurements difficult or QTc data uninterpretable
   5. history of additional risk factors for torsades de pointe (eg, heart failure, hypokalemia, family history of long QT syndrome).
9. History of alcoholism or drug/chemical abuse.
10. Alcohol consumption of >14 units (females) and >21 units (males) per week. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
11. Positive alcohol breath test result or positive urine drug screen, including cotinine (confirmed by repeat) at screening or check in.
12. Positive hepatitis panel and/or positive human immunodeficiency virus test.
13. Any of the following haematology values at screening or check-in, as confirmed by 1 repeat if necessary:

    1. haemoglobin <11 g/dL for females, and <12 g/dL for males
    2. absolute neutrophil count <1.5 × 109/L (<1500/µL).
14. Renal or liver impairment at screening or check-in defined as, confirmed by 1 repeat if necessary:

    1. serum creatinine ≥135 µmol/L
    2. ALT and/or AST ≥2 × ULN
    3. ALP and/or total bilirubin >1.5 × ULN (an isolated total bilirubin >1.5 × ULN is acceptable if total bilirubin is fractionated and direct bilirubin is <35%).
15. Participation in a clinical study involving administration of an investigational drug (new chemical entity) or medical device within the last 90 days or 5 half-lives of the investigational medication, whichever is longer, prior to dosing.
16. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing.
17. Use or intend to use any prescription medications/products within 14 days or 5 half lives of the medication/product, whichever is longer, prior to check-in (hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives are acceptable).
18. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 14 days prior to check in.
19. Use or intend to use slow release medications/products considered to still be active within 14 days prior to check in.
20. Received live attenuated vaccination within 6 weeks prior to screening or intends to receive such a vaccination during the study.
21. Use of tobacco or nicotine containing products (including but not limited to; cigarettes, electronic cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum) within 6 months prior to check-in and the inability to abstain from nicotine-containing products until the follow-up visit.
22. Receipt of blood products within 2 months prior to check in.
23. Donation of blood (>400 mL) or comparable blood loss (>350 mL) from 3 months prior to screening, plasma donation from 2 weeks prior to screening, or platelets donation from 6 weeks prior to screening.
24. Poor peripheral venous access.
25. Consumption of caffeine-containing foods and beverages within 72 hours of screening or is unable to abstain from caffeine-containing foods and beverages from 7 days prior to check in until discharge.
26. Consumption of any foods or beverages which alter CYP1A2 activity, eg, barbecued food or cruciferous vegetables, such as broccoli and cauliflower, within 14 days prior to check-in (a list of prohibited foods will be provided to subjects).
27. Consumption of any foods or beverages containing Seville-type oranges, grapefruit, or poppy seeds within 7 days prior to check-in.
28. Have previously completed or withdrawn from this study, and have previously received the IMP.
29. Subjects who, in the opinion of the investigator (or designee; including input from subjects' general practitioner, as applicable), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Number of treatment related adverse event, including abnormal laboratory events | Day -1 to follow up (7-14 days after discharge)
  All AEs, including clinical laboratory, vitals signs, body temperature, respiratory rate, physical examinations and ECGs will be analyzed in all subjects receiving HTL0014242

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose
  The observed peak plasma concentration determined from the plasma
Area under the curve (AUC) from time 0 to 24 hours postdose (AUC0-24h) | predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose
  Area under the plasma concentration-time curve up to 24h
time to reach the maximum observed plasma concentration (tmax) | predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose
  time to reach the maximum observed plasma concentration (tmax)
Area under the curve (AUC) from time 0 to the time of the last quantifiable concentration (AUC0-tlast) | predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose
  Area under the plasma concentration-time curve up to the last measurable timepoint
Area under the curve (AUC) from time 0 extrapolated to infinity (AUC0-∞) | predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose
  Area under the curve, calculated as AUC0-tlast + C0-tlast/λz, where C0-tlast is the last observed measurable concentration
t1/2 and kel | predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose
  apparent initial elimination half-life (t1/2) and associated elimination rate onstant (kel)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, PhD, Principal Investigator — Covance; Hamzah Malik, Study Director — Covance; Robert Holland, BMBCh, DPhil, Study Director — Heptares Therapeutics Ltd
Locations (1):
- Covance, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No